CLINICAL TRIAL: NCT01607749
Title: Asthma Educational Intervention on Physical Education Teachers in Primary Schools
Brief Title: Study for Asthma Education in Primary Schools
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Manuel Praena-Crespo, MD, Head Researcher Pediatrics, Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GESA
Record Dates: First submitted 2011-11-23; First posted 2012-05-30 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Asthma
Keywords: Asthma Control; Quality of life; Children; Asthma education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational Program (Experimental): Students in the intervention schools learn the educational program "Asthma, Sport and Health" in three sessions during a period of 6 weeks. The content of the educational program has been published elsewhere.
  Interventions: Behavioral: Educational Program
- Asthma information for teachers (No Intervention): Information about asthma the Ministry of Education to all schools in the community.
  Interventions: Other: Usual Asthma Information for teachers

INTERVENTIONS:
Behavioral: Educational Program — Schools in the intervention group received the educational program "Asthma, Sport and Health", as validated by our group. This program will be taught to students in three lessons with equipment designed and developed by the research group to be taught within the curriculum of physical education subject.
  Teachers of physical education specialists responsible for the project at each center will receive the training curriculum for use in a training seminar for a school day by researchers from the health of our group. Once familiar with the educational package of three sessions taught his students and fellow faculty (on different days for teachers and students) within 15-30 days.
  Arms: Educational Program
Other: Usual Asthma Information for teachers — Common asthma information for teachers
  Arms: Asthma information for teachers

SUMMARY:
Undertake a study of educational intervention in primary schools in Andalusia

HYPOTHESIS:

There are differences in quality of life associated with asthma (as measured by the questionnaire PAQLQ) and the level of asthma control in students with asthma aged 11 and 12 years who receive an educational intervention with their peers without asthma versus those receiving standard information in schools.

OBJECTIVES: To compare the control of asthma symptoms, quality of life in asthma and asthma knowledge among a group receiving an educational intervention delivered by specialist teachers of physical education (MEEF) in Primary Schools (CEIP) and control.

MÉTODOS group: Randomized controlled single-blind.

POPULATION: Students of 11 and 12 years old in Andalusia

Sample size: 258 children / children with asthma for a mean contrast (alpha error of 3.4%. 80% power, a confidence level of 95% considering 20% loss. 2580 students will be enrolled prevalence of asthma 10%) . Conglomerates of the CEIP in urban, rural, public and private-reached.

INTERVENTION: Training MEEF with the educational program "Sports and Health Asthma and subsequent delivery, then the students MEEF are 5th and 6th grade ( 3 sessions). CONTROL: The standard instruction in schools. OUTCOME VARIABLES: Quality of life (Juniper) and "control del asthma en niños"(CAN) in asthmatics, Knowledge (NAKQ questionnaire) and attitudes toward asthma (all students and teachers). Pre-intervention (T0), post-intervention at 5-6 months (T1)

Independent variables: Sex, suffering or not asthma, intervention / control, type CEIP.

STATISTICAL ANALYSIS: Comparison of continuous variables: T Students (If normal distribution) "Mann-Whitney (If non-normal distribution). To study qualitative variables chi-square test (normal distribution) and Kruskal-Wallis ( no-normal distribution).

DETAILED DESCRIPTION:
DESIGN. Single-blind clinical trial with random allocation to the group receiving educational intervention and control group, developed throughout the school year (September 2011 to May 2012). The unit of randomization will be the schools to avoid intracenter contamination of the students during the educational intervention. The units of analysis are the students of schools FIELD OF STUDY. Students aged 10 and 13 years old attending school and Primary Education (CEIP) in Andalusia, a world population of 38,829 students from a total of 728 CEIP. The schools will be recruited through AVERROES tool of the Ministry of Education of the Andalusia

Sample size:

To achieve a power of 90.0% to detect differences in the contrast of the null hypothesis H ₀: μ ₀ = μ ₀ by t-Student test bilaterally for two independent samples, considering that the significance level is 5%, and assuming a mean difference to the quality of life questionnaire between groups of 0.5 and the common standard deviation is 1.10 units, with estimated losses of 15% is necessary to include 129 units in the experimental group Reference and 129 units in the Experimental group, totaling 258 experimental units in the study. Since the prevalence of asthma is approximately 10% in our population, we need to include a total of 2580 students, for a total of 258 students with asthma and other students will be students without asthma who get the outcome measures and compare your average asthma knowledge and attitudes to asthma of all students involved in the study and teaching centers.

INVITATION TO PARTICIPATE:

CEIP will be chosen by randomization by computer, which will be offered to participate. One of the researchers contacted the directors and teachers of Physical Education (MEF) of the sites, explaining the purpose of the study. Upon acceptance to participate, seek the approval of the School Councils to inform parents of students about the study, again requesting consent for their children's participation in the trial.

ASSIGNMENT randomly to two groups:

The allocation will be 1:1 in the control group and intervention group, after school stratification by public / private and rural / urban, by number of students enrolled in schools will be invited to participate. (Annex 1) As for the post randomisation losses, estimated at 15%, for not attending educational sessions at 3 is an analysis by intention to treat and per protocol. In those subjects lost to follow up and can be reached, apply them to complete the study questionnaires and PAQLQ ACT to determine the degree of asthma control and quality of life before the completion of the course. Randomization to intervention and control centers shall be made to avoid contamination between control and intervention that occur within a single center.

Blinding:

The research team will train in the use of educational package to the MEF will be different from the group of researchers who collected the questionnaires, the questionnaires correction made without knowing which group was assigned to the student and therefore do not know the type of intervention in the CES. Teachers and students in the intervention and control groups did not examine the content of the curriculum of another comparison group. The researchers who conducted the statistical treatment, will not know the assignment to experimental and control centers will have a key for identification. The Principal Investigator will know the allocation of control and experimental groups

Intervention:

Schools in the intervention group received the educational program "Asthma, Sport and Health" 23, as validated by our grupo24 to be taught within the curriculum of the CEIP once you have been approved by the school board for each center. This program will be taught to students in three lessons with equipment designed and developed by the research group to be taught within the curriculum of the CEIP. The contents of each class and its methods of work are detailed in the same educational program. However it offers a framework in Annex 2.

Teachers of physical education specialists responsible for the project at each center will receive the training curriculum for use in a training seminar for a school day by researchers from the health of our group. Once familiar with the educational package of three sessions taught his students and fellow faculty (on different days for teachers and students) within 15-30 days.

CONTROL: The control group provides information on asthma that supplies the Ministry of Education to all schools in the community.

STUDY VARIABLES:

For the main hypothesis "An intervention through an educational program to all students, with or without asthma in primary schools can improve the quality of life associated with asthma (as measured by the questionnaire PQALQ) and level of asthma control (measured with the questionnaire ACT) and students with asthma, "the study variables are:

• Dependent variable (primary):

* Level of quality of life achieved through the following: (PAQLQ). Quantitative values ranging between 1 and 7. The minimal clinically important difference is 0.5 points.

  * The level of asthma control achieved during follow-up. and "control del asthma en niños"(CAN) in asthmatics: Quantitative values ranging between 5 and 25. The minimal clinically important difference is 3.7 points.
  * Dependent Variable (secondary objective)
* Knowledge of asthma with the questionnaire NAKQ. Quantitative values ranging between 0 and 31.
* Attitudes towards asthma among teachers and students, between the intervention and control. We will use a questionnaire based on a model that includes multiple domains (internal control, tolerance to asthma, chance and external control) detailed in ANNEX 5. Is filled following a Liker scale between 1 and 6 strongly agree strongly disagree.
* Measures to protect asthmatics applied in primary schools after the educational intervention on students and faculty obtained by researchers in schools. Quantitative values ranging between 0 and 20 (ANNEX 7)

PERFORMANCE MEASUREMENT TOOLS:

1. Quality of Life Questionnaire in children with asthma-version with standardized activities (PAQLQ (S) of E. Juniper, validated Spanish. (Consists of 23 items with values for poorer quality of life 1, best value 7 per item, which are averaged together) APPENDIX 3
2. Control of asthma (ACT). Annex 4
3. asthma knowledge questionnaire will use the asthma knowledge questionnaire of Newcastle, whose linguistic validation was conducted by our group and approved by their original authors. ANNEX 5. This questionnaire has a maximum score of 31, with a range of possible values between 0-31.
4. Survey of attitudes to asthma. We will use a questionnaire based on a model that includes multiple domains (internal control, tolerance to asthma, chance and external control) detailed in ANNEX 6. Is filled following a Liker scale between 1 and 6 strongly agree strongly disagree.
5. Resource Questionnaire Asthma at School (Annex 7)
6. Data Sheet for students with authorization for treatment in case of crisis. Baseline questionnaires were used for measuring and monitoring quality of life, asthma control, attitudes to asthma knowledge questionnaire on asthma and asthma Resources at CES. The questionnaires were obtained before surgery (T0), and 6 months after it (T1) to check the duration of the changes obtained after intervention.

DATA ANALYSIS:

At baseline, we intergroup comparison (intervention and control) of qualitative variables using the chi-square test or Fisher's exact test when necessary. Quantitative variables follow or not as a normal distribution (Shapiro Wilks test) were analyzed with Student's t-or Mann-Whitney, respectively.

In the mean intragroup comparison (intervention or control) repeated throughout the study, apply the Student t-test for related samples Wilcoxon or in the event of non-normality. To compare means of the 2 study groups during follow-up will use repeated measures ANOVA on the assumption of normality and the assumption of non-normality in each group will discuss any changes with the Wilcoxon test.

The analysis was performed using SPSS-V18. Analysis by intention to treat: They take into account the results for each group initially assigned, regardless of the intervention, to meet the program's effectiveness in real conditions.

There will also be a per protocol analysis to determine the effectiveness of the program in ideal conditions.

DIFFICULTIES AND LIMITATIONS OF THE STUDY:

1. Selection bias. In the case of children with asthma are not included in the study all children who may have asthma, or by the refusal to know or because the disease is diagnosed in many cases and is only recognized by euphemistic terms . Randomization could solve the problem between intervention and control
2. Losses.

   * Refusal by the parents of patients selected to participate in the study.
   * Lack of cooperation throughout the study by faculty and / or students.
   * We have chosen a large enough sample for the study lacks statistical power no.
   * provide for losses in the entire study from the first randomization of the sample universe.
   * Change of school that the student belongs. 3) You may bias awareness of the subjects included in the study by the mere fact of knowing and not being observed strict consequence of the educational intervention. Random assignment of intervention and control groups minimize their influence.

     4) Intervention studies with training activities, increase the level of knowledge of pathology addressed, but do not always produce positive changes in attitudes aimed at controlling the disease.

ethical

1. The project has been approved by the Ethics Committee for Health Research Health District Primary Care Sevilla dated April 15, 2009. (ANNEX 9)
2. After completing the study, the primary schools involved in the control arm receive the same treatment as the intervention group
3. Parents will be obtained informed consent
4. Confidentiality of data. The information contained herein is

ELIGIBILITY:
Inclusion Criteria:

* Studying in fifth and sixth year of primary education

Exclusion Criteria:

* Intellectual deficit to answer questions.
* Do not to sign the parent informed consent

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4506 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 months
  We measure the quality of life through the Pediatric Asthma Quality of Life Questionnaire (Elizabeth Juniper)
Asthma Control | 6 months

SECONDARY OUTCOMES:
Measurement of attitudes toward asthma | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Praena-Crespo, PhD, Principal Investigator — Centro de Salud La Candelaria. Sevilla. Servicio Andaluz de Salud
Locations (2):
- Spain (2):
  - Centro de Salud La Candelaria, Seville, Andalusia
  - Universidad Pablo de Olavide, Seville, Andalusia

REFERENCES:
- [Derived] Praena-Crespo M, Aquino-Llinares N, Fernandez-Truan JC, Castro-Gomez L, Segovia-Ferrera C; GESA network. Asthma education taught by physical education teachers at grade schools: A randomised cluster trial. Allergol Immunopathol (Madr). 2017 Jul-Aug;45(4):375-386. doi: 10.1016/j.aller.2016.10.022. Epub 2017 Mar 18. PMID 28318759